COORDINATE Informed consent form V 2.1 Edited 02.11.2022

## APPENDIX B INFORMED CONSENT FORM

## **COORDINATE**

CRP fOr respiratORy DIagnosis iN Kyrgyz pediATric practicE









## **Appendix B** Informed Consent Participant's Identification Number Date (DD/MM/YYYY) Study site n years months Age Read the following statement to the parent/caregiver. "Hello. I am\_\_\_\_\_\_, I am a member of the COORDINATE Project team. I am here with my colleagues to study the problem of respiratory diseases and irrational prescription of antibiotics to children. I would like to observe to your child consultation by a healthcare worker at this medical center. Your child may have capillary blood drawn from the ring finger for a Creactive protein test to clarify the diagnosis and evaluate the severity of the disease. Your child will be examined and treated even if you choose not to have your child involved. Rest assured that the information will be kept confidential and you can withdraw your child's participation at any time or refrain from answering any questions." "At this time, do you want to ask me anything about this?" "Do I have your agreement to participate?" Name of child: Date: Phone number: Signature:\_\_\_\_